CLINICAL TRIAL: NCT06559644
Title: Assessment of the Safety and Efficacy of Hema-NeoTIL01 Cell Infusion Therapy in Relapsed/Refractory Acute Leukemia: A Single-Arm, Open-Label, Prospective Study
Brief Title: Hema-NeoTIL01 Cell Infusion Therapy in Relapsed/Refractory Acute Leukemia
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Hema-NeoTIL01-SU01
Record Dates: First submitted 2024-05-14; First posted 2024-08-19 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-05

CONDITIONS: Leukemia, Myeloid, Acute; B-cell Acute Lymphoblastic Leukemia
Keywords: B-ALL; AML; T cell therapy
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Burkitt Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hema-NeoTIL01 treatment (Experimental): In this study, we adopted a 3+3 design with dose escalation. Initially, three dose groups were established: 2.0×10^7, 6.0×10^7, and 2.0×10^8 cells/kg. Each dose group received treatment on Days 0, 3, and 6 through i.v. injection, with bone marrow examination performed on Day 7 to assess tumor burden. Upon assessment by the investigators and discussion with the Safety Review Committee (SRC), it will be determined that whether patients may benefit from additional infusions. With SRC approval, the number of administrations could be increased, not exceeding a maximum of six doses. At the end of dose escalation, the SRC may decide to adjust the number of participants in the designated dose group as deemed appropriate.
  Interventions: Biological: Hema-NeoTIL01

INTERVENTIONS:
Biological: Hema-NeoTIL01 — Patients will receive intravenous infusion of Hema-NeoTIL01, which is a highly specific tumor infiltrating lymphocyte (TIL) product derived from patients' bone marrow or peripheral blood, expanded ex vivo through antigen presentation.

SUMMARY:
This clinical trial aims to investigate the safety, optimal dosage, and effectiveness of autologous tumor-specific T cells, known as Hema-NeoTIL0 in treating relapsed/refractory B-ALL/AML.

DETAILED DESCRIPTION:
Primary Objective:

To assess the safety of Hema-NeoTIL01 in the treatment of relapsed/refractory acute leukemia (B-ALL/AML).

Secondary Objective:

To evaluate the efficacy of Hema-NeoTIL01 in relapsed/refractory acute leukemia (B-ALL/AML).

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 and <70 years old, gender not specified;
2. Diagnosed with B-ALL or AML according to the World Health Organization (WHO) classification of hematopoietic and lymphoid tissue tumors (2022 version);
3. Meet the diagnosis of relapsed/refractory leukemia, excluding isolated extramedullary relapse; For relapsed or refractory ALL, including any of the following situations: a) Relapse: Peripheral blood or bone marrow recurrence of primitive cells >5% or extramedullary lesions appear again after complete remission; b) Refractory: Primary refractory patients who fail to achieve complete remission after standard induction chemotherapy; Or meet the diagnosis of relapsed or refractory AML, including any of the following situations: a) Relapse: Recurrence of primitive cells >5% in bone marrow after complete remission (except for reasons such as bone marrow regeneration after consolidation chemotherapy) or extramedullary infiltration of leukemia cells; b) Refractory: Patients who have failed two cycles of standard treatment; those who relapse within 12 months after CR after consolidation therapy; those who relapse after 12 months and are ineffective after conventional chemotherapy; those with two or more relapses; those with persistent extramedullary leukemia;
4. Patients who have previously received ineffective/relapsed CAR-T cell therapy may be included in this study, provided that the efficacy evaluation of CAR-T therapy has been completed and evaluated as NR, or relapse after remission of CAR-T therapy;
5. Estimated survival >12 weeks;
6. Eastern Cooperative Oncology Group (ECOG) performance status score ≤2;
7. Left ventricular ejection fraction (LVEF) ≥50%;
8. Pulmonary function ≤Grade 1 dyspnea (CTCAE v5.0), normal oxygen saturation without oxygen supplementation;
9. Total bilirubin (TBil) ≤3×upper limit of normal (ULN), aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤5×ULN, creatinine ≤1.6mg/dL;
10. Pregnancy test must be negative, and fertile non-abstinent female patients must agree to use effective contraception from the start of self-screening to 1 year after cell infusion. Fertile male patients with fertile partners must agree to use effective contraception from the start of self-screening to 1 year after cell infusion, and should not donate semen or sperm throughout the study period.
11. The subject and their legal guardian voluntarily participate in this study, understand the trial information and objectives, and provide informed consent with a signed and dated signature.
12. The subject and their legal guardian are willing and able to comply with all trial requirements.

Exclusion Criteria:

1. Patients with a history of severe central nervous system diseases, such as uncontrolled seizures, stroke, severe brain injury resulting in aphasia, paralysis, dementia, Parkinson's disease, psychiatric disorders, etc.;
2. New York Heart Association (NYHA) functional class III or IV heart failure;
3. Any unstable diseases occurring within 6 months before screening (including but not limited to): unstable angina, ischemic or cerebrovascular accidents, myocardial infarction, severe arrhythmias requiring drug treatment (such as rapid atrial fibrillation, high-degree atrioventricular block, ventricular tachycardia, ventricular fibrillation, or torsades de pointes), cardiac catheterization or coronary artery stenting, or coronary artery bypass surgery, thrombotic or embolic events.
4. Presence of disseminated intravascular coagulation;
5. Severe autoimmune diseases or immunodeficiency diseases;
6. Active graft-versus-host disease requiring continued systemic therapy;
7. Subjects receiving systemic corticosteroids or other immunosuppressive therapy before screening, and the investigator determines that they will continue to use long-term therapy after enrollment (excluding inhalation or local use);
8. History of or concomitant active malignant tumors, excluding cured non-invasive basal cell or squamous cell skin cancer, uterine cervical carcinoma in situ or localized prostate cancer or breast ductal carcinoma in situ without recurrence for at least 2 years;
9. Presence of other severe medical conditions as determined by the investigator, such as uncontrolled hypertension or diabetes, severe renal insufficiency, severe pulmonary dysfunction, etc.;
10. Active HBV or HCV infection (HBV-DNA positive or HCV-RNA positive), HIV positive, or syphilis positive;
11. Other severe or persistent active infections;
12. Severity of adverse events related to previous systemic immunotherapy (including other investigational drugs or medical device interventions) at screening not reduced to grade 1 or baseline status;
13. Discontinuation of immunosuppressants within 2 weeks prior to screening;
14. History of allergy to any component of the cell product;
15. Vaccination or any surgical procedure within 4 weeks prior to screening;
16. Other conditions deemed by the investigator to potentially increase subject risk or interfere with trial results.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
CR/CRi, MRD-negative CR | Within 28 days after the first dose
  Complete remission (CR) is defined as the presence of less than 5% bone marrow blasts in an aspirate containing spicules, accompanied by independence from transfusions.
  CR with incomplete hematologic recovery (CRi) is defined as the presence of less than 5% bone marrow blasts, with either an absolute neutrophil count (ANC) of less than 1×10^9/L or a platelet count of less than 100×10^9/L, while remaining transfusion-independent but exhibiting persistent cytopenia.
  Minimal residual disease (MRD)-negative CR is defined as a leukemic cell count below the sensitivity threshold of 1×10^-4 (0.01%) of bone marrow mononuclear cells (MNCs), as measured by multiparameter flow cytometry.

SECONDARY OUTCOMES:
RFS | 2 years
  Relapse-free survival (RFS) is defined as the interval from the date of achieving CR to the first occurrence of leukemia relapse, death, or the date of the last follow-up.
OS | 2 years
  Overall survival (OS) is defined as the duration from the time of enrollment to death from any cause.
Adverse events | Within 28 days after the first dose
  The number of adverse events are evaluated with CTCAE V5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaowen Tang, Study Chair — The First Affiliated Hospital of Soochow University
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No